CLINICAL TRIAL: NCT00488189
Title: Association of Antibiotic Utilization Measures and Control of Extended-Spectrum β-Lactamases (ESBLs) Producing Bacteria
Brief Title: Study Evaluation Tazocin Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0910X-102370
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2010-06

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Piperacillin, Tazobactam Drug Combination; Piperacillin; Tazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): baseline, collecting rectal swab samples
- 2 (Active Comparator): use pipercill/tazobact to replace 3rd generation cephalosporin and collect rectal swab
  Interventions: Drug: Tazocin (pipercillin/tazobactam)

INTERVENTIONS:
Drug: Tazocin (pipercillin/tazobactam) — over 50% third generation cephalosporin should be replaced by Pip/Taz
  Arms: 2

SUMMARY:
This is an antibiotic intervention study to determine the value of using piperacillin/tazobactam in reducing the cases of ESBL producing E. coli or K. pneumoniae colonization and infection.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted or transferred to ICU/Pulmonary units
* Patients of either sex, 18 years of age or older

Exclusion Criteria:

- Patients who stay in units less than 48 hours will not be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
1. The acquisition rate of ESBL producing E. coli or K. Pneumoniae at the end of phase I (pre-intervention) and phase II (last 3 months of intervention phase) | 9 months

SECONDARY OUTCOMES:
The infection rate due to ESBL producing E. coli or K. pnumoniae at the end of phase I (pre-intervention) and phase II (last 3 months of intervention phase) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For China, medinfo@wyeth.com
Locations (1):
- Beijing, Beijing Municipality, China